CLINICAL TRIAL: NCT00395174
Title: Comparison of the Immunogenicity, Safety and Reactogenicity of FluBlok, Trivalent Recombinant Baculovirus-Expressed Hemagglutinin Influenza Vaccine, to a Licensed Egg-Grown Influenza Vaccine In Ambulatory Elderly Adults
Brief Title: Comparison of the Immunogenicity, Safety and Reactogenicity of FluBlok, To a Licensed Vaccine In Elderly Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Manon Cox, Chief Operating Officer, Protein Sciences Corporation
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PSC03
Record Dates: First submitted 2006-10-30; First posted 2006-11-02 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluBlok

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FluBlok (Experimental): Recombinant Trivalent Hemagglutinin Influenza Vaccine: 2005-2006 formulation containing 45μg of each hemagglutinin derived from A/New Caledonia (H1N1), A/Wisconsin (H3N2) and B/Ohio
  135μg total
  Interventions: Biological: Influenza Vaccination
- TIV (Fluzone) (Active Comparator): Licensed trivalent influenza vaccine (TIV): 2005-2006 formulation containing 15μg of each hemagglutinin derived from A/Wisconsin (H3N2), A/New Caledonia (H1N1) and B/Malaysia
  45μg total
  (Fluzone, sanofi pasteur)
  Interventions: Biological: Influenza Vaccination

INTERVENTIONS:
Biological: Influenza Vaccination — 0.5mL dose for intramuscular injection
  Other Names: FluBlok; Fluzone; rHA; rHA0; recombinant hemagglutinin; TIV

SUMMARY:
The purpose of this study were to obtain additional evidence in support of the safety and immunogenicity of a recombinant hemagglutinin (rHA) vaccine in an elderly population, and to establish non-inferiority of the immunogenicity of the rHA vaccine when compared with a licensed trivalent influenza vaccine (TIV). Another purpose was to provide a preliminary estimate of the relative efficacy of the two vaccines against culture-positive influenza-like illness during the subsequent epidemic.

DETAILED DESCRIPTION:
Annual influenza epidemics are associated with serious excess morbidity and mortality, particularly among the elderly. Licensed trivalent inactivated influenza vaccines (TIVs) have been shown to reduce hospitalization and death following influenza in this vulnerable population, but their efficacy is lower than that observed in younger, healthy populations. In addition, recent studies have questioned the level of effectiveness of TIV in the elderly, suggesting that cohort studies have overestimated the benefits of immunization with current TIV formulations in this age group. In view of these considerations, it is widely accepted that improved and alternative vaccines are needed for control of seasonal and pandemic influenza.

Currently available TIVs are prepared from viruses that are grown in embryonated hens' eggs. Alternative substrates for vaccine production are desirable in order to reduce the vulnerability of and to expand influenza vaccine supply. Recombinant DNA techniques allow for expression of the influenza hemagglutinin (rHA) by baculovirus vectors in insect cell cultures. Advantages of this technique include speed of production, absence of egg protein, and a highly purified product. Previous studies among healthy younger and older adults have confirmed that rHA vaccines are safe, well tolerated and immunogenic at dosages up to nine times higher than those contained in TIV. Dose-related increases in serum antibody levels after immunization also were observed.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adults aged 65 and older
* Medically stable, as determined by oral temperature <100.0°F, medical history, and targeted physical examination based on medical history
* Able to understand and comply with planned study procedures
* Provides written informed consent prior to initiation of any study procedure.

Exclusion Criteria:

* Known allergy to eggs or other vaccine components.
* Immunosuppression as a result of an underlying illness or treatment, or used anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Any malignancy (excluding nonmelanotic skin cancer or lymphoproliferative disorder), other than localized prostrate cancer, diagnosed or treated actively during the past 5 years. Subjects with any history of lymphoproliferative disorder will be excluded, while subjects with a history of localized nonmelanotic skin cancer may be eligible.
* Long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids within the preceding 6 months (Nasal and topical steroids are allowed).
* Major psychiatric diagnosis including schizophrenia, bipolar disease or other major depression, or any diagnosis of dementia or associated concomitant medications (e.g., Aricept) used for treating dementia
* History of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Receipt of any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* History of severe reactions following immunization with influenza virus vaccines.
* Moderate to severe acute illness or febrile illness (oral temperature greater than 100*F) within 1 week prior to vaccination.
* Receipt of an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during study period.
* Known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* History of alcohol or drug abuse in the last 5 years.
* History of Guillain-Barré Syndrome.
* Any acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, interfere with the evaluation of responses, or render the subject unable to meet the requirements of the protocol. These conditions include, but are not limited to: history of significant renal impairment (dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease); subjects with diabetes mellitus, well-controlled with oral agents may enroll as long there has been no dosage increase within the past 6 months; insulin-dependent diabetes is excluded; cardiac insufficiency, if heart failure is present (New York Heart Association Functional Class III or IV); an arteriosclerotic event during the 6 months prior to enrollment (e.g., history of myocardial infarction, stroke, recanalization of femoral arteries, or transient ischemic attack).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 870 (Actual)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and reactogenicity of FluBlok and TIV in medically stable adults 65 years and older. | influenza season

SECONDARY OUTCOMES:
Comparison of relative efficacy and effectiveness of FluBlok and TIV in medically stable adults 65 years and older. | influenza season
Evaluation and comparison of immunogenicity of FluBlok and TIV in medically stable adults 65 years and older. | influenza season

CONTACTS AND LOCATIONS:
Overall Officials: Wendy A. Keitel, MD, Principal Investigator — Baylor College of Medicine; Hana M. El-Sahly, MD, Principal Investigator — Baylor College of Medicine; John J. Treanor, MD, Principal Investigator — University of Rochester Medical; Keith S. Reisinger, MD, Principal Investigator — Primary Physicians research; Gregory A. Poland, MD, Principal Investigator — Mayo Clinic College of Medicine; Kenneth D. Lessans, MD, Principal Investigator — Passport Health Maryland; John J. Minneti, MD, Principal Investigator — Passport Health New Jersey; Kristen Lyke, MD, Principal Investigator — Center of Vaccine Development, University of Maryland
Locations (7):
- United States (7):
  - Center of Vaccine Development, Univ. of Maryland, Baltimore, Maryland
  - Passport Health Maryland, Baltimore, Maryland
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Passport Health New Jersey, Shrewsbury, New Jersey
  - Rochester Medical Center, Rochester, New York
  - Primary Physicians Research, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Keitel WA, Treanor JJ, El Sahly HM, Gilbert A, Meyer AL, Patriarca PA, Cox MM. Comparative immunogenicity of recombinant influenza hemagglutinin (rHA) and trivalent inactivated vaccine (TIV) among persons > or =65 years old. Vaccine. 2009 Dec 11;28(2):379-85. doi: 10.1016/j.vaccine.2009.10.037. Epub 2009 Oct 29. PMID 19879222
- [Derived] Rajendran M, Nachbagauer R, Ermler ME, Bunduc P, Amanat F, Izikson R, Cox M, Palese P, Eichelberger M, Krammer F. Analysis of Anti-Influenza Virus Neuraminidase Antibodies in Children, Adults, and the Elderly by ELISA and Enzyme Inhibition: Evidence for Original Antigenic Sin. mBio. 2017 Mar 21;8(2):e02281-16. doi: 10.1128/mBio.02281-16. PMID 28325769
- [Derived] Nachbagauer R, Choi A, Izikson R, Cox MM, Palese P, Krammer F. Age Dependence and Isotype Specificity of Influenza Virus Hemagglutinin Stalk-Reactive Antibodies in Humans. mBio. 2016 Jan 19;7(1):e01996-15. doi: 10.1128/mBio.01996-15. PMID 26787832
- See also: Related Info — http://proteinsciences.com